CLINICAL TRIAL: NCT05746923
Title: Lesser Poland Cracovian Heart Failure Registry
Acronym: LECRA-HF
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Konrad Stępień, MD, Jagiellonian University
Other Study IDs: 1072.6120.349.2022
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Heart Failure Acute
Keywords: heart failure; acute heart failure; decompensation; revascularization; long-term prognosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LECRA-HF patients: The study population consists of hospitalized patients with acute heart failure who are over 18 years of age, both women and men. Patients will be initially categorized into one of three groups based on the current European Society of Cardiology (ESC) heart failure guidelines based on left ventricular ejection fraction (LVEF) values: patients with reduced (LVEF ≤40%), mildly reduced (LVEF 41-49%) and preserved (LVEF ≥50%) ejection fraction.

SUMMARY:
The goal of Lesser Poland Cracovian Heart Failure Registry (LECRA-HF) is to expand the knowledge about acute heart failure (AHF) and its long-term prognosis.

The main questions are:

* assessment of long-term prognosis of AHF and its determinants
* determination of the optimal AHF treatment methods
* assessment of indications for invasive coronary arteries diagnostics and revascularization and their long-term effects
* analysis of the particular HF subtypes (HFimpEF, HFpEF, HFsnEF, HFrEF, HFmrEF)

DETAILED DESCRIPTION:
LECRA-HF is a registry of patients with acute heart failure (AHF) hospitalized in the Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow, Jagiellonian University Medical College. So far, a small population of patients has been included in similar registries conducted in the Polish population. This did not allow to draw reliable conclusions about this diverse group of patients.

As part of the LECRA-HF registry, a comprehensive analysis of the clinical characteristics of patients is planned, taking into account their medical history, anthropometric measurements, results of electrocardiographic, imaging and laboratory tests, as well as the treatment used during the index hospitalization and after discharge. Their long-term prognosis will also be analyzed. LECRA-HF is a continuous registry, updated annually until 2026.

The data collected in the LECRA-HF will be used to distinguish and describe relatively new subtypes of HF (HFimpEF, HFsnEF) as well as to properly characterize that difficult and very diverse population with a serious long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization due to acute heart failure
* > 18 years of age

Exclusion Criteria:

* inability to give informed consent to participate in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of hospitalized patients with acute heart failure who are over 18 years of age, both women and men. Patients will be initially categorized into one of three groups based on the current European Society of Cardiology (ESC) heart failure guidelines based on left ventricular ejection fraction (LVEF) values: patients with reduced (LVEF ≤40%), mildly reduced (LVEF 41-49%) and preserved (LVEF ≥50%) ejection fraction.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  Mortality due to all causes

SECONDARY OUTCOMES:
Cardiovascular mortality | 2 years
  Mortality due to CV causes
HF rehospitalizations | 2 years
  Rehospitalizations related to HF decompensation

OTHER OUTCOMES:
LVEF increase >10% in the follow-up echocardiography | 2 years
  In accordance with HFimpEF definition

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Nessler, Prof., Study Chair — Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow; Konrad Stępień, MD, Principal Investigator — Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow
Locations (1):
- Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow, Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No